CLINICAL TRIAL: NCT00838162
Title: A Phase IIa, Open-label, Randomized Trial in Treatment-naive HIV-1-infected Subjects to Determine the Antiviral Activity of 14 Days of Monotherapy With 4 Different Dose Regimens of TMC310911 Coadministered With Ritonavir
Brief Title: A Study to Determine the Antiviral Activity of TMC310911 When Administered With Ritonavir in Treatment-Naive Human Immunodeficiency Virus - Type 1 (HIV-1) Infected Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR015952; TMC310911-TIDP21-C201 (Other: Tibotec Pharmaceuticals, Ireland); 2008-008190-58 (EudraCT Number)
Record Dates: First submitted 2009-02-05; First posted 2009-02-06 (Estimated); Results first posted 2013-03-07 (Estimated); Last update posted 2013-06-12 (Estimated); Status verified 2013-06

CONDITIONS: Human Immunodeficiency Virus Type 1
Keywords: Human immunodeficiency virus type 1; HIV-1; HIV-1 treatment-naive; TMC310911; Protease inhibitor; Ritonavir; Antiviral Activity; HIV Infections; Treatment Naive
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections | interventions — TMC-310911; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- TMC310911/rtv 75/100 mg twice daily (Experimental): TMC310911 75 mg + ritonavir 100 mg twice daily on Days 1 to 14
  Interventions: Drug: TMC310911 75 mg twice daily; Drug: Ritonavir 100 mg twice daily
- TMC310911/rtv 150/100 mg twice daily (Experimental): TMC310911 150 mg + ritonavir 100 mg twice daily on Days 1 to 14
  Interventions: Drug: TMC310911 150 mg twice daily; Drug: Ritonavir 100 mg twice daily
- TMC310911/rtv 300/100 mg twice daily (Experimental): TMC310911 300 mg + ritonavir 100 mg twice daily on Days 1 to 14
  Interventions: Drug: TMC310911 300 mg twice daily; Drug: Ritonavir 100 mg twice daily
- TMC310911/rtv 300/100 mg once daily (Experimental): TMC310911 300 mg + ritonavir 100 mg once daily on Days 1 to 14
  Interventions: Drug: TMC310911 300 mg once daily; Drug: Ritonavir 100 mg once daily

INTERVENTIONS:
Drug: TMC310911 75 mg twice daily — TMC310911 75 mg twice daily orally (by mouth) on Days 1 to 14.
  Arms: TMC310911/rtv 75/100 mg twice daily
Drug: TMC310911 150 mg twice daily — TMC310911 150 mg twice daily orally (by mouth) on Days 1 to 14
  Arms: TMC310911/rtv 150/100 mg twice daily
Drug: TMC310911 300 mg twice daily — TMC310911 300 mg twice daily orally (by mouth) on Days 1 to 14
  Arms: TMC310911/rtv 300/100 mg twice daily
Drug: TMC310911 300 mg once daily — TMC310911 300 mg once daily orally (by mouth) on Days 1 to 14
  Arms: TMC310911/rtv 300/100 mg once daily
Drug: Ritonavir 100 mg twice daily — Ritonavir 100 mg twice daily orally (by mouth) on Days 1 to 14
  Arms: TMC310911/rtv 150/100 mg twice daily; TMC310911/rtv 300/100 mg twice daily; TMC310911/rtv 75/100 mg twice daily
Drug: Ritonavir 100 mg once daily — Ritonavir 100 mg once daily orally (by mouth) on Days 1 to 14
  Arms: TMC310911/rtv 300/100 mg once daily

SUMMARY:
The purpose of this study is to evaluate the antiviral activity as measured by the change in viral load from baseline in the 14 days following initiation of treatment with 4 different dose regimens of TMC310911 co-administered with ritonavir.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention) and randomized (study medication assigned by chance) study in treatment-naive human immunodeficiency virus type 1 (HIV-1)-infected participants (participants who had not been treated with a therapeutic HIV vaccine within 1 year prior to enrollment and who had never been treated with an antiretroviral [ARV] medication indicated for the treatment of HIV-infection or ARVs for treatment of hepatitis B infection with anti-HIV activity prior to screening). In this study approximately 32 participants will be enrolled and randomly assigned to receive 4 different dose regimens co-administered with ritonavir (8 participants in each dosing regimen). The trial will consist of a screening period (maximum 6 weeks), a treatment period with TMC310911 (2 weeks), and a follow-up period (4 weeks). Safety evaluation will include assessment of adverse events, clinical laboratory tests, vital sign measurements, physical examinations and electrocardiograms.

ELIGIBILITY:
Inclusion Criteria:

* Documented human immunodeficiency virus type 1 (HIV-1) infection for at least 6 months prior to the screening date
* Participant who has not been treated with a therapeutic HIV vaccine within 1 year prior to enrolment and has never been treated with an antiretroviral (ARV) medication indicated for the treatment of HIV infection or ARVs for treatment of hepatitis B-infection with anti-HIV activity
* Participant agrees not to start antiretroviral therapy (ART) before the baseline visit
* Able to comply with the protocol requirements and have good accessible veins
* HIV-1 plasma viral load at screening visit of above 5,000 HIV-1 Ribonucleic acid copies/mL
* CD4+ cell count above 200 cells/mm3 at screening

Exclusion Criteria:

* HIV-2 infected participants and/or participants with any active or chronic hepato-renal disease
* Life expectancy of less than 6 months
* Documented acute (primary) HIV-1 infection
* Pre-existing protease inhibitor (PI) medication resistance
* Any currently active Acquired Immunodeficiency Syndrome (AIDS) - defining illness
* Any active clinically significant disease or findings during screening or medical history or physical examination that in the investigator's opinion, would compromise the outcome of the study
* Any confirmed grade 3 or 4 toxicity according to the Division of AIDS (DAIDS) grading scale at screening

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2009-06; Primary Completion 2009-08 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals, Ireland Clinical Trial, Study Director — Tibotec Pharmaceuticals, Ireland
Locations (3):
- Germany (3):
  - Berlin
  - Frankfurt
  - Hamburg

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in Germany.
Pre-assignment Details: In total, 41 participants were screened of whom 33 participants were randomized and treated with TMC310911. All treated participants completed the study; there were no dropouts or discontinuations during the study.
Groups:
- TMC310911/Rtv 300/100 mg Once a Day: TMC310911 300 mg + ritonavir 100 mg once a day on Days 1 to 14
Period: Overall Study
Arm/Group | TMC310911/Rtv 75/100 mg Twice Daily | TMC310911/Rtv 150/100 mg Twice Daily | TMC310911/Rtv 300/100 mg Twice Daily | TMC310911/Rtv 300/100 mg Once a Day
Started | 9 | 8 | 8 | 8
Completed | 9 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TMC310911/Rtv 75/100 mg Twice Daily | TMC310911/Rtv 150/100 mg Twice Daily | TMC310911/Rtv 300/100 mg Twice Daily | TMC310911/Rtv 300/100 mg Once a Day | Total
Number analyzed (Participants) | 9 | 8 | 8 | 8 | 33
Age Continuous [Mean (Standard Deviation); unit: years] | 29.7 (7.23) | 38.1 (8.66) | 35.5 (6.87) | 37.8 (10.19) | 35.1 (8.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 0 | 0 | 1
  Male | 8 | 8 | 8 | 8 | 32
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 8 | 8 | 8 | 8 | 32
  Black | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Changes From Baseline in Plasma log10 Human Immunodeficiency Virus Type 1 Ribonucleic Acid (HIV-1 RNA)
Description: The antiviral activity of TMC310911 is measured by the change in viral load from baseline in the 14 days of treatment following initiation of treatment with 4 different dosing regimens of TMC310911 coadministered with ritonavir.
Time Frame: Baseline (Day 1), Day 8, Day 15
Population: Intent-to treat (ITT) population- participants who received at least 1 dose of study medication (TMC310911).
Measure: Mean (Standard Error); unit: log10 copies/mL
Arm/Group | TMC310911/Rtv 75/100 mg Twice Daily | TMC310911/Rtv 150/100 mg Twice Daily | TMC310911/Rtv 300/100 mg Twice Daily | TMC310911/Rtv 300/100 mg Once a Day
Number analyzed (Participants) | 9 | 8 | 8 | 8
log10 copies/mL
  Baseline | 4.72 (0.245) | 4.36 (0.259) | 4.78 (0.161) | 4.71 (0.116)
  Day 8 | -1.30 (0.126) | -1.14 (0.147) | -1.07 (0.104) | -1.06 (0.144)
  Day 15 | -1.53 (0.117) | -1.79 (0.192) | -1.69 (0.103) | -1.55 (0.160)

2. Secondary Outcome: Number of Participants With Virologic Response at Any Timepoint During the 14-day Treatment Period
Description: Virologic response is a viral load test result below a chosen threshold value (less than 50 copies/mL, less than 400 copies/mL, or at least 1 log drop in viral load) at any timepoint during a 14-day treatment of 4 different dose regimens of TMC310911 coadministered with 100 mg ritonavir.
Time Frame: 14 days
Population: Intent-to-treat (ITT) Population- all randomized participants who received at least 1 dose of study medication (TMC310911)
Measure: Number; unit: Participants
Arm/Group | TMC310911/Rtv 75/100 mg Twice Daily | TMC310911/Rtv 150/100 mg Twice Daily | TMC310911/Rtv 300/100 mg Twice Daily | TMC310911/Rtv 300/100 mg Once a Day
Number analyzed (Participants) | 9 | 8 | 8 | 8
Participants
  Viral load less than 50 copies/mL | 0 | 1 | 0 | 0
  Viral load less than 400 copies/mL | 3 | 4 | 1 | 0
  At least 1 log10 Viral Load Drop | 9 | 8 | 8 | 7

3. Secondary Outcome: Mean Changes From Baseline in CD4+ Cell Count
Time Frame: Baseline (Day 1), Day 8, Day 15
Population: Intent-to-treat (ITT) Population - all randomized participants who received at least 1 dose of study medication (TMC310911)
Measure: Mean (Standard Error); unit: x 1000000 cells/L
Arm/Group | TMC310911/Rtv 75/100 mg Twice Daily | TMC310911/Rtv 150/100 mg Twice Daily | TMC310911/Rtv 300/100 mg Twice Daily | TMC310911/Rtv 300/100 mg Once a Day
Number analyzed (Participants) | 9 | 8 | 8 | 8
x 1000000 cells/L
  Baseline | 575.7 (56.97) | 464.9 (61.32) | 494.0 (70.43) | 479.6 (39.16)
  Day 8 | -21.0 (41.23) | 40.3 (45.19) | -14.8 (47.59) | 17.9 (48.20)
  Day 15 | -33.7 (27.04) | -2.8 (31.44) | -2.0 (41.23) | 92.5 (58.70)

4. Secondary Outcome: Maximum Plasma Concentration (Cmax) of TMC310911
Time Frame: Day 1 and Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | TMC310911/Rtv 75/100 mg Twice Daily | TMC310911/Rtv 150/100 mg Twice Daily | TMC310911/Rtv 300/100 mg Twice Daily | TMC310911/Rtv 300/100 mg Once a Day
Number analyzed (Participants) | 9 | 8 | 8 | 8
ng/mL
  Day 1 | 487.9 (450.3) | 623.0 (358.1) | 706.3 (553.2) | 1924 (1048)
  Day 14 | 589.7 (554.1) | 1674 (652.3) | 2256 (961.9) | 2963 (1920)

5. Secondary Outcome: Time to Reach the Maximum Plasma Concentration (Tmax) of TMC310911
Time Frame: Day 1 and Day 14
Population: as for outcome 3
Measure: Median (Full Range); unit: hours
Arm/Group | TMC310911/Rtv 75/100 mg Twice Daily | TMC310911/Rtv 150/100 mg Twice Daily | TMC310911/Rtv 300/100 mg Twice Daily | TMC310911/Rtv 300/100 mg Once a Day
Number analyzed (Participants) | 9 | 8 | 8 | 8
hours
  Day 1 | 5.02 [2.00 to 12.00] | 5.00 [3.00 to 8.12] | 5.06 [5.00 to 12.17] | 5.00 [2.00 to 5.02]
  Day 14 | 4.98 [1.00 to 8.00] | 3.00 [1.00 to 5.03] | 3.87 [0.00 to 5.02] | 3.02 [1.02 to 5.03]

6. Secondary Outcome: Area Under the Plasma Concentration-time Curve (AUC12) From the Time of Administration of TMC310911 up to 12 Hours After Dosing
Time Frame: Day 1 and Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | TMC310911/Rtv 75/100 mg Twice Daily | TMC310911/Rtv 150/100 mg Twice Daily | TMC310911/Rtv 300/100 mg Twice Daily | TMC310911/Rtv 300/100 mg Once a Day
Number analyzed (Participants) | 8 | 8 | 7 | 7
ng.h/mL
  Day 1 | 2519 (2123) | 2735 (1572) | 2990 (2245) | 10040 (6122)
  Day 14 | 4031 (3845) | 10680 (3147) | 16010 (8229) | 17520 (11610)

7. Secondary Outcome: Predose Plasma Concentration (C0h) of TMC310911
Time Frame: Day 2, Day 3, Day 4, Day 6, Day 8, Day 10, Day 12 and Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | TMC310911/Rtv 75/100 mg Twice Daily | TMC310911/Rtv 150/100 mg Twice Daily | TMC310911/Rtv 300/100 mg Twice Daily | TMC310911/Rtv 300/100 mg Once a Day
Number analyzed (Participants) | 9 | 8 | 8 | 8
ng/mL
  Day 2 | 79.95 (104.1) | 207.7 (122.9) | 231.9 (199.9) | 45.48 (28.94)
  Day 3 | 93.98 (92.90) | 448.0 (266.1) | 586.3 (454.2) | 125.9 (69.01)
  Day 4 | 88.94 (113.6) | 291.3 (170.2) | 1035 (552.2) | 191.0 (175.7)
  Day 6 | 119.1 (182.1) | 443.0 (284.7) | 960.5 (506.9) | 250.0 (236.1)
  Day 8 | 134.5 (179.0) | 665.9 (461.1) | 1028 (724.1) | 239.6 (242.6)
  Day 10 | 78.51 (57.88) | 394.4 (134.4) | 736.1 (435.0) | 251.7 (211.0)
  Day 12 | 104.6 (82.91) | 518.6 (288.7) | 1110 (547.5) | 250.2 (181.9)
  Day 14 | 152.5 (248.2) | 420.9 (244.6) | 924.8 (527.9) | 209.9 (187.2)

8. Secondary Outcome: Average Steady-state Plasma Concentration (Css,av) of TMC310911
Time Frame: Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | TMC310911/Rtv 75/100 mg Twice Daily | TMC310911/Rtv 150/100 mg Twice Daily | TMC310911/Rtv 300/100 mg Twice Daily | TMC310911/Rtv 300/100 mg Once a Day
Number analyzed (Participants) | 8 | 7 | 7 | 8
ng/mL | 336.2 (321.3) | 889.6 (262.6) | 1340 (689.6) | 887.3 (567.5)

9. Secondary Outcome: Fluctuation Index of TMC310911
Description: Fluctuation index, ie, percentage fluctuation: variation between maximum (Cmax) and minimum (Cmin) plasma concentration at steady-state, calculated as: 100 x ([Cmax-Cmin]/Css,av). Css,av is an average steady-state plasma concentration.
Time Frame: Day 14
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percent ng/mL
Arm/Group | TMC310911/Rtv 75/100 mg Twice Daily | TMC310911/Rtv 150/100 mg Twice Daily | TMC310911/Rtv 300/100 mg Twice Daily | TMC310911/Rtv 300/100 mg Once a Day
Number analyzed (Participants) | 8 | 7 | 7 | 8
Percent ng/mL | 181.0 (80.00) | 161.3 (29.22) | 129.2 (52.89) | 331.8 (55.47)

ADVERSE EVENTS:
Time Frame: Up to 4 weeks after the last dose administration of study medication
Arm/Group | TMC310911/Rtv 75/100 mg Twice Daily | TMC310911/Rtv 150/100 mg Twice Daily | TMC310911/Rtv 300/100 mg Twice Daily | TMC310911/Rtv 300/100 mg Once a Day
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 5/9 | 5/8 | 6/8 | 3/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TMC310911/Rtv 75/100 mg Twice Daily (N=9) | TMC310911/Rtv 150/100 mg Twice Daily (N=8) | TMC310911/Rtv 300/100 mg Twice Daily (N=8) | TMC310911/Rtv 300/100 mg Once a Day (N=8)
Conjunctivitis (Eye disorders) | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abnormal faeces (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 3 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Discomfort (General disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 3 | 2 | 4 | 0
Influenza like illness (General disorders) | 1 | 0 | 0 | 0
Cytomegalovirus hepatitis (Infections and infestations) | 0 | 0 | 0 | 1
Folliculitis (Infections and infestations) | 0 | 1 | 0 | 0
Genital herpes (Infections and infestations) | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Skeletal injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 1
Micturition urgency (Renal and urinary disorders) | 2 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days